CLINICAL TRIAL: NCT04899466
Title: A Prospective Study Evaluating the Efficacy of ActiGraft in Secondary Closure of Abdominal Surgical Wound Dehiscence
Brief Title: Efficacy Evaluation of ActiGraft in Secondary Closure of Abdominal Surgical Wound Dehiscence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RedDress Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD008
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Dehiscence Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ActiGraft (Experimental): Whole blood clot (WBC) gel
  Interventions: Device: ActiGraft

INTERVENTIONS:
Device: ActiGraft — Whole blood clot (WBC) gel

SUMMARY:
This is a prospective, single arm study, consisting of 20 women with abdominal surgical wound dehiscence that requires secondary closure. The participants will receive a weekly application of ActiGraft for 4 weeks, or until complete healing of the wound (the earlier of the two).

An historic matched-control group of 20 patients will be compared retrospectively

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Women that had a laparotomy no more than 3 weeks before accrual.
* Surgical wound dehiscence that requires a secondary closure.
* Time from wound dehiscence >24 hours and <6 days.
* The open wound includes epidermis, dermis and sub cutaneous fat.
* The patient can sign an informed consent form.

Exclusion Criteria:

* Patients with necrotizing fasciitis
* Patients with fascial dehiscence
* Cannot withdraw blood in the required amount (up to 18 mL per week).
* Known coagulation problems, abnormal thrombocytes level or if heparin is given intravenously. Subjects who are taking oral anti-coagulants or anti-agreganrts will not be excluded.
* Pregnancy
* Subject is currently receiving (i.e., within the past 30 days) or scheduled to receive systemic steroids (Prednisone- more than 10mg/d or equivalent).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of complete wound closure | 4 weeks
  Skin re-epithelialization without drainage or dressing requirements

SECONDARY OUTCOMES:
Wound Percent Area Reduction (PAR) | 2, 4 and 6 weeks
  The change in wound area (decrease or increase) with respect to the area at baseline, expressed as a percentage.
Mean time of complete wound closure | 4 weeks
  Skin re-epithelialization without drainage or dressing requirements
Durability of wound closure 2 weeks after complete healing | Up to 6 weeks
  No wound dehiscence
Comparison of time to complete closure between study cases and historic control | 4 weeks
  Skin re-epithelialization without drainage or dressing requirements

OTHER OUTCOMES:
Change in pain level | 1, 2, 3 and 4 weeks
  Measured by Numeric Rating Scale (0 - no pain at all to 10 - worst pain) weekly for 4 weeks post ActiGraft application
Patient satisfaction | 1, 2, 3, 4, 6 weeks and 42 days
  Will be assessed by subject satisfaction survey using a 5-point Likert Scale (the higher score means a better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Sirota, Study Director — RedDress Ltd.
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: Yes
The results will be part of several scientific publications
Supporting Information: Study Protocol
Time Frame: Upon publication